CLINICAL TRIAL: NCT00846430
Title: Medical Treatment of "High-Risk" Neurofibromas in Patients With Type 1 Neurofibromatosis: A Clinical Trial of Sequential Medical Therapies
Brief Title: Medical Treatment of "High-Risk" Neurofibromas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Albert Cornelius, MD, Corewell Health West
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-260; 2008-260 (Other: Spectrum Health)
Record Dates: First submitted 2009-01-16; First posted 2009-02-18 (Estimated); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Neurofibromatosis 1
Keywords: Neurofibromas; Neurofibromatosis 1; Celecoxib; Celebrex; Peg-Interferon alpha-2b; PEG-Intron; Temozolomide; Temodar; Vincristine Sulfate; Oncovin
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma | interventions — peginterferon alfa-2b; Celecoxib; Temozolomide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label Intervention (Experimental): This is a phase II single arm study with sequential treatments available by response where all participants begin therapy with a combination of celecoxib and interferon alpha-2b (CI, treatment-1). Response to CI therapy will be assessed at six months by clinical and radiographic evaluations. Those patients who have achieved a partial response (improvement in pain, improvement in functioning, or ≥50% reduction in tumor size) or complete response (resolution of pain, and normalization of functioning with a ≥ 90% reduction in tumor size) will continue with the same CI therapy for up-to two years on study.
  Interventions: Drug: Peg-Interferon alpha-2b; Drug: Celecoxib (Celebrex); Drug: Temozolomide (temodar); Drug: Vincristine Sulfate (Oncovin)

INTERVENTIONS:
Drug: Peg-Interferon alpha-2b — age and weight dependant
Drug: Celecoxib (Celebrex) — age and weight dependant
Drug: Temozolomide (temodar) — age and weight dependant
Drug: Vincristine Sulfate (Oncovin) — age and weight dependant

SUMMARY:
Patients with neurofibromatosis type 1 (NF1) commonly develop non-cancerous tumors called plexiform neurofibromas. These tumors can be defined as "high-risk" when they result in severe pain, physical disability, organ dysfunction and/or become life-threatening. Presently, there is no effective medical therapy to offer patients with "high-risk" plexiform neurofibromas, and surgery does not provide lasting help. This study will evaluate the effectiveness of two treatment combinations in patients with "high-risk" plexiform neurofibromas.

DETAILED DESCRIPTION:
The study's design involves treating eligible patients with a combination of celecoxib and pegylated interferon alpha-2b. If the patients have at least a partial response after six months, they may continue on the same treatment for up to two years. If the patient experiences less than a partial response, or has progressive disease after six months of therapy, then vincristine and temozolomide will be added to the celecoxib and interferon alpha-2b backbone. Response to treatment will be assessed after a minimum of six months, presuming the patient has not experienced progressive disease. Total duration of therapy on study is two years for any individual treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* "High-Risk" Plexiform Neurofibromas associated with a diagnosis of NF1
* 2-30 years old (minimum bodyweight of 10 kilograms)
* Adequate renal function

Exclusion Criteria:

* Previously untreated active optic glioma
* History of any previous allergy to study medications
* History of ischemic vascular disease
* Pregnancy / Breast feeding

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert S Cornelius, MD, Principal Investigator — Helen DeVos Children's Hospital
Locations (1):
- Helen DeVos Children's Hospital, Grand Rapids, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Period 1: Baseline to 6 months", "Period 2: After 6 month evaluation for addition of vincristine and temozolomide", if accurate and appropriate
Period: Overall Study
Arm/Group | Open-Label Intervention
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label Intervention
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Symptoms and Pain
Description: Subjects will be evaluated for pain and Quality of Life scores
Time Frame: Monthly physical exam first three months and then every three months after, for up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Intervention
Number analyzed (Participants) | 9
Participants | 9

2. Primary Outcome: At Least 50% Shrinkage in Tumor Measurements by Physical Examination
Time Frame: Monthly physical exam first three months and then every three months after, for up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Intervention
Number analyzed (Participants) | 9
Participants | 7

3. Primary Outcome: Response by MRI Measurements
Description: partial response by RICST criteria is defined as >50% tumor shrinkage
Time Frame: evaluated 6, 12 and 24 months compared to baseline
Measure: Number; unit: participants
Arm/Group | Open-Label Intervention
Number analyzed (Participants) | 9
participants
  Partial Response at 6 months | 0
  Complete Response at 6 months | 1
  Less than Partial Response at 6 months | 8
  Partial Response at 12 months | 2
  Complete Response at 12 months | 1
  Less than Partial Response at 12 months | 6
  Partial Response at 24 months | 4
  Complete Response at 24 months | 1
  Less than Partial Response at 24 months | 1
  no longer participating at 24 months | 3

4. Secondary Outcome: No Reported Psychological Toxicity Based Upon Psychological Evaluations
Description: Psychological toxicity defined as suicidal ideation
Time Frame: Psychological evaluation at 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Intervention
Number analyzed (Participants) | 9
Participants | 8

ADVERSE EVENTS:
Time Frame: collected over 5 years
Description: adverse events collected during provider appointments
Arm/Group | Open-Label Intervention
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Intervention (N=9)
Suicidal Ideation (Psychiatric disorders) | 1 (1) — hospitalized for suicidal ideation, expected side effect of interferon.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Intervention (N=9)
Fatigue (Nervous system disorders) | 1 (1) — difficulty maintaining school attendance

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-06-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT00846430/Prot_SAP_000.pdf